CLINICAL TRIAL: NCT00955266
Title: A Randomized Double-Blind Placebo-Controlled Trial of Intravenous Calcium and Myocardial Diastolic Dysfunction During Separation From Cardiopulmonary Bypass
Brief Title: A Trial of Intravenous Calcium and Myocardial Diastolic Dysfunction During Separation From Cardiopulmonary Bypass
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Michael Nurok, MD, PhD, Cardiac Anesthesiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009-P-000052
Record Dates: First submitted 2009-07-30; First posted 2009-08-10 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Diastolic Dysfunction
Keywords: Separation; Cardiopulmonary bypass; Calcium chloride
MeSH Terms: interventions — Calcium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calcium Chloride (Active Comparator): Calcium chloride, 10mg/kg
  Interventions: Drug: Calcium Chloride
- Placebo (Placebo Comparator): Normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcium Chloride — Calcium chloride 10mg/kg in 50cc NS delivered over 5 minutes
  Arms: Calcium Chloride
Drug: Placebo — Normal saline, 50cc delivered over 5 minutes
  Arms: Placebo

SUMMARY:
Successful heart surgery requires the resumption of a strong beating heart prior to separation from the heart and lung machine. There are different ways to do this. At this hospital, the surgical team usually gives calcium to people when they come off of the heart and lung machine because some doctors believe that calcium can "jump start" the heart. Not every hospital does this.

Some people think that calcium may have a side effect of making the heart more stiff. Stiff hearts do not beat as well or receive as much blood to tissues as non-stiff hearts. If calcium makes the heart stiff, then doctors may have to use other medicines to support the heart in the operating room and the intensive care unit. This may ultimately lead to poorer outcomes including a longer stay in the intensive care unit and in the hospital.

This study is being performed to find out if calcium has the side effect of making the heart more stiff. This study compares calcium to placebo. The placebo looks exactly like the calcium, but it contains no calcium. During this study patients may receive placebo instead of calcium. Neither the doctor nor the study team will know which drug the subject will receive.

ELIGIBILITY:
Inclusion Criteria:

* Men and women greater than 18 years of age
* Undergoing primary elective valve surgery at Brigham and Women's Hospital
* Consented for Transesophogeal Echocardiography (TEE) as part of routine intra-operative care and monitoring

Exclusion Criteria:

* Patients not consented for TEE as part of routine intra-operative care
* Any absolute contraindication to TEE
* Ionized calcium level < 0.80 mmol/L near separation from CPB
* Myocardial infarction (MI) or acute coronary syndromes < 3 months prior to surgery due to the presence of pre-operative diastolic dysfunction in infarcted or ischemic myocardium
* Ejection fraction (EF) < 35%
* Atrial fibrillation / flutter the absence of an A wave on mitral inflow Doppler
* Heart rate (HR) > 100 during 2 data point collections due to E / A wave superimposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Nurok, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Womens Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcium Choloride: Calcium chloride, 10mg/kg
  Calcium Chloride: Calcium chloride 10mg/kg in 50cc NS delivered over 5 minutes
Period: Overall Study
Arm/Group | Calcium Choloride | Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcium Choloride | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Diastolic Dysfunction
Description: E/ A ratio on TEE. This ratio of peak velocity flow in early diastole (the E wave) to peak velocity flow in late diastole caused by atrial contraction (the A wave) is reflective of degree of diastolic dysfunction.
Time Frame: 64 enrolled patients or 9 months following start of protocol, whichever comes first
Population: Data was in paper form only. Data storage location sustained significant water intrusion and mold contamination in June 2016. Environmental contractor has advised paper contents will need to be destroyed under containment conditions to ensure that mold does not spread. As a result, data is not available for results reporting.
Arm/Group | Calcium Choloride | Placebo
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

2. Secondary Outcome: Return to Cardiopulmonary Bypass Secondary to Hemodynamic Instability
Description: Return to Cardiopulmonary bypass Yes/ No
Time Frame: 64 enrolled patients or 9 months following start of protocol, whichever comes first
Population: as for outcome 1
Arm/Group | Calcium Choloride | Placebo
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

3. Secondary Outcome: Need for Inotropic or Vasopressor Support Upon Leaving the OR
Description: Use of inotropes or vasopressors in the Operating Room.
Time Frame: 64 enrolled patients or 9 months following start of protocol, whichever comes first
Population: as for outcome 1
Arm/Group | Calcium Choloride | Placebo
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

4. Secondary Outcome: Length of Hospital Stay (Days)
Description: Hospital length of stay in days.
Time Frame: 64 enrolled patients or 9 months following start of protocol, whichever comes first
Population: as for outcome 1
Arm/Group | Calcium Choloride | Placebo
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

5. Secondary Outcome: Length of ICU Stay (Days)
Description: Intensive Care Unit length of stay in days.
Time Frame: 64 enrolled patients or 9 months following start of protocol, whichever comes first
Population: as for outcome 1
Arm/Group | Calcium Choloride | Placebo
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year.
Arm/Group | Calcium Choloride | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
Data storage location sustained significant water intrusion and mold contamination in June 2016. Environmental contractor has advised contents of location need to be destroyed. As a result, data is not available for results reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes